CLINICAL TRIAL: NCT04931628
Title: Efficacy and Safety of Salvianolic Acid on Acute Ischemic Stroke
Brief Title: Efficacy and Safety of Salvianolic Acid on AIS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: negative information
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: First Affiliated Hospital of Wenzhou Medical University (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Zhejiang University (Other); Ningbo No. 1 Hospital (Other); Zhejiang Hospital (Other); Zhejiang Provincial Tongde Hospital (Other); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); Xiaoshan People's Hospital (Other); Red Cross Hospital, Hangzhou, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-092
Record Dates: First submitted 2021-06-14; First posted 2021-06-18 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Stroke
Keywords: Stroke, ischemic, Acute
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — salvianolic acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- salvianolic acid group (Active Comparator): salvianolic acid group 100mg+0.9%NaCl 250ml, injection, 14 days
  Interventions: Drug: Salvianolic Acid
- 0.9% NaCl (Placebo Comparator): 0.9%NaCl 250ml, injection, 14 days
  Interventions: Drug: 0.9% NaCl

INTERVENTIONS:
Drug: Salvianolic Acid — salvianolic acid, injection, 100mg+0.9%NaCl 250ml, qd, 14 days
  Arms: salvianolic acid group
Drug: 0.9% NaCl — 0.9% NaCl
  Arms: 0.9% NaCl

SUMMARY:
Stroke has the characteristics of high morbidity, disability and fatality rate, which brings heavy spiritual and economic burdens to the family, society and the country. In my country, 33%-50% of ischemic strokes are attributed to intracranial atherosclerosis.

Studies have shown that oxidative stress, increased blood viscosity, and damage to vascular endothelial cells are important mechanisms for the development of cerebral infarction. Salvia miltiorrhiza is a commonly used traditional Chinese medicine in traditional medicine in my country. Salvia miltiorrhiza polyphenolic acid is the effective ingredient of salvia miltiorrhiza. It is the water-soluble active part of salvia miltiorrhiza. It can resist oxidation, anticoagulation, antiplatelet, cell protection, and expand blood vessels, thereby achieving protection Cardiovascular system.

The purpose of this study was to evaluate the effects and adverse effects of salvianolic acid on acute ischemic stroke onset within 72 hours, and to evaluate the improvement of patients' ischemic area perfusion and clinical function scores.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke with the first onset, or a history of cerebral infarction but with a modified Rankin Scale (mRS) score ≤1, onset within 72h;
2. CT examination to rule out cerebral hemorrhage;
3. With clear signs of nervous system positioning, the National Institutes of Health Stroke Scale (NIHSS) score ≥ 4

Exclusion Criteria:

1. Diseases with bleeding tendency;
2. Liver and kidney dysfunction;
3. Malignant tumors or those undergoing anti-tumor treatment;
4. Allergic physique, allergic to aspirin or Salvianolic Acid;
5. Heart failure, multiple system failure;
6. Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
MRS score | 90 days
  MRS score ≤2

SECONDARY OUTCOMES:
Cerebral blood flow volume (CBV) | 90 days
  Cerebral blood flow volume
Cerebral blood flow (CBF) | 90 days
  Cerebral blood flow
NIHSS score | 90 days
  NIHSS score
Adverse drug reactions (ADR) | 90 days
  Adverse drug reactions

CONTACTS AND LOCATIONS:
Locations (1):
- Dai Haibin, Hangzhou, Zhejiang, China